CLINICAL TRIAL: NCT06450457
Title: Effects of High Intensity Stepping Training on Gait in Patients With Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kaitlin Benjamin, Student, Principal Investigator, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MH-23-1064
Record Dates: First submitted 2024-05-29; First posted 2024-06-10 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- High intensity stepping program (Experimental): The high intensity stepping training consists of a one-hour long physical therapy session administered by a physical therapist, and it will include overground walking, treadmill walking (with or without bodyweight support), stairs, and resisted walking. Heart rate will be monitored with the Polar heart rate monitor, with the goal of reaching moderate to high intensity for 30 minutes during the one hour-long physical therapy session. The training may involve the use of the Therastride Treadmill System or the VECTOR Bioness, and the device used will be determined by how much assistance the participant needs. If a participant is already ambulating and doesn't need assistance, then that participant won't use any equipment other than a Polar heart rate monitor.
  Interventions: Device: Polar H10 heart rate monitor; Device: Therastride Treadmill System; Device: VECTOR Bioness; Other: Physical therapy

INTERVENTIONS:
Device: Polar H10 heart rate monitor — Heart rate will be monitored using a Polar H10 heart rate monitor, with the goal of reaching moderate to high intensity for 30 minutes during the one hour long therapy intervention.
Device: Therastride Treadmill System — Participants will be asked to walk on the Therastride Treadmill for 30 minutes.This treadmill can unweight patients so that the task of walking becomes easier. The body weight can be adjusted depending on how much assistance a patient needs from 0% of their bodyweight (completely independent) to up to 50% of their bodyweight for the purposes of this study.
Device: VECTOR Bioness — Participants will be asked to walk using the VECTOR Bioness on a track outside the gym with a harness attached to an overhead sling system. This system can unweight patients so that the task of walking becomes easier. The body weight can be adjusted depending on how much assistance a patient needs from 0% of their bodyweight (completely independent) to up to 50% of their bodyweight for the purposes of this study. This system allows for overground walking on a small indoor track as opposed to walking on a treadmill.
Other: Physical therapy — Physical therapy will be administered by a physical therapist and will include overground walking, treadmill walking, stairs, and resisted walking.

SUMMARY:
The purpose of this study is to examine the effects of high intensity stepping training on gait recovery, including walking speed and endurance, in patients with cerebellar ataxia. The hypothesis is that there will be a significant improvement in gait outcome measures (6 Minute Walk Test and 10 Meter Walk Test) in patients who receive high-intensity stepping training during physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ataxia
* admitted to The Institute for Rehabilitation and Research (TIRR) Texas Medical Center (TMC) Inpatient or TIRR Kirby Glenn Outpatient
* pathology that primarily affects the brain/cerebellum, including degenerative diseases, stroke, traumatic brain injury (TBI), posterior fossa tumor, and multiple sclerosis (MS)
* ambulatory at initial evaluation or will have functional ambulation goals at initial evaluation (as noted by 10 meter walk test and 6 minute walk test measures documented as 0)
* chronicity of injury will be of at least 1 month or greater

Exclusion Criteria:

* diagnoses that may have cerebellar involvement but without cerebellar ataxia as a principal impairment such as autism, down syndrome, schizophrenia, etc
* non ambulatory or who are not able to participate in high intensity stepping training due to cardiac involvement (such as cardiac rehabilitation parameters) or due to orthopedic limitations (such as weight bearing parameters)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlin Benjamin, PT, DPT, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Intensity Stepping Program: The high intensity stepping training consists of a 1-hour long physical therapy session administered by a physical therapist, and it will include overground walking, treadmill walking (with or without bodyweight support), stairs, and resisted walking. Heart rate will be monitored with the Polar heart rate monitor, with the goal of reaching moderate to high intensity for 30 minutes during the one hour-long physical therapy session. The training may involve the use of the Therastride Treadmill System or the VECTOR Bioness, and the device used will be determined by how much assistance the participant needs. If a participant is already ambulating and doesn't need assistance, then that participant won't use any equipment other than a Polar heart rate monitor.
  Therastride Treadmill System: Participants will walk on the Therastride Treadmill for 30 minutes. This treadmill can unweight patients so that the task of walking becomes easier. Body weight can be adjusted depending on how much assistance a patient needs from 0% of their bodyweight (completely independent) to up to 50% of their bodyweight.
  VECTOR Bioness: Participants will walk using the VECTOR Bioness on a track outside the gym with a harness attached to an overhead sling system. Body weight can be adjusted depending on how much assistance a patient needs from 0% of their bodyweight (completely independent) to up to 50% of their bodyweight. This system allows for overground walking on a small indoor track.
Period: Overall Study
Arm/Group | High Intensity Stepping Program
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High Intensity Stepping Program
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 58.75 [41 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Walking Speed in Meters Per Second as Assessed by the 10 Meter Walk Test(10MWT)
Description: Participant is asked to walk a distance of 10 meters and the speed is measured by dividing the distance covered by the time taken.
Time Frame: Baseline, 3 weeks
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | High Intensity Stepping Program
Number analyzed (Participants) | 4
meters per second
  Baseline | 0.13 (0.16)
  3 weeks | 0.60 (0.31)

2. Primary Outcome: Distance Walked in Feet as Assessed by the the Six Minute Walking Test (6MWT)
Description: Participants will be asked to walk as far as possible for 6 minutes. Longer distance walked shows better outcome.
Time Frame: Baseline, 3 weeks
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | High Intensity Stepping Program
Number analyzed (Participants) | 4
feet
  Baseline | 145.26 (177.34)
  3 weeks | 423.10 (260.55)

3. Secondary Outcome: Ataxia as Assessed by the Scale for the Assessment and Rating of Ataxia (SARA)
Description: Scale for the Assessment and Rating of Ataxia (SARA) measures ataxia with a total score that ranges from 0 (no ataxia) to 40 (most severe ataxia). A higher score indicates a worse outcome.
Time Frame: Baseline, 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stepping Program
Number analyzed (Participants) | 4
score on a scale
  Baseline | 25.25 (7.80)
  3 weeks | 17.87 (9.15)

4. Secondary Outcome: Ability to Balance as Assessed by the Berg Balance Scale (BBS)
Description: Berg Balance Scale measures balance with a total score that ranges from 0 to 56. A higher score indicates better balance.
Time Frame: Baseline, 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Intensity Stepping Program
Number analyzed (Participants) | 4
score on a scale
  Baseline | 9.50 (13.22)
  3 weeks | 20.00 (16.18)

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Arm/Group | High Intensity Stepping Program
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT06450457/Prot_SAP_000.pdf